CLINICAL TRIAL: NCT05914155
Title: The Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rituximab (Genetical Recombination) for the Treatment for Idiopathic Membranous Nephropathy with Nephrotic Syndrome （PRIME Study）
Brief Title: Clinical Study of Rituximab for the Treatment for Idiopathic Membranous Nephropathy with Nephrotic Syndrome
Acronym: PRIME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shoichi Maruyama MD PhD (Other)
Responsible Party: Sponsor-Investigator, Shoichi Maruyama MD PhD, Professor, Nagoya University
Organization: Nagoya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAMCR-020
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Glomerulonephritis, Membranous; Nephrotic Syndrome，Idiopathic
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrosis, Lipoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rituximab group in double-blind phase (Active Comparator)
  Interventions: Drug: Rituximab (genetical recombination)
- Placebo group in double-blind phase (Placebo Comparator)
  Interventions: Drug: Placebo
- Rituximab group in open-label phase (Other)
  Interventions: Drug: Rituximab (genetical recombination)

INTERVENTIONS:
Drug: Rituximab (genetical recombination) — Administer 1,000 mg of rituximab (genetical recombination) IV infusion every two weeks for two doses in double-blind phase.
  Arms: Rituximab group in double-blind phase
Drug: Placebo — Administer placebo IV infusion every two weeks for two doses in double-blind phase.
  Arms: Placebo group in double-blind phase
Drug: Rituximab (genetical recombination) — Patients who remain to be ICR II (Incomplete Remission Type II) or NR (No Response) until Week 26 in the double-blind phase, if the patients wish to move to the open-label phase and the investigator or a subinvestigator considers the move necessary, the patient will move to the open-label phase and receive 1,000 mg of rituximab (genetical recombination) IV infusion every two weeks for two doses after the readministration criteria are confirmed to be met.
  Arms: Rituximab group in open-label phase

SUMMARY:
To confirm the efficacy and safety of rituximab (genetical recombination) intravenously administered to idiopathic membranous nephropathy with nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo kidney biopsy and are diagnosed as having idiopathic membranous nephropathy prior to the obtainment of informed consent
2. Patients who are diagnosed as having nephrotic syndrome prior to the obtainment of informed consent and receive no steroids or immunosuppressants within 12 weeks prior to the obtainment of informed consent
3. Patients with urine protein-creatinine ratio ≥ 3.5 g/gCr at the screening
4. Patients with hypoalbuminemia (serum albumin ≤ 3.0 g/dL) at the screening
5. Patients aged 15 years or older at informed consent
6. Patients who give voluntary written consent after having received adequate information on this study (legally acceptable representatives should also give consent for underage patients, and informed assent should be obtained from children)

Exclusion Criteria:

1. Patients with primary nephrotic syndrome other than membranous nephropathy (IgA nephropathy, minimal change disease, focal segmental glomerulosclerosis and so forth), and patients with secondary nephrotic syndrome (autoimmune disease, metabolic disease, infection, allergic/hypersensitive disease, tumor, and drug-induced disease)
2. Patients with the renal function lowered (eGFR <30 mL/min/1.73 m2 based on CKD-EPIcr formula) at the screening
3. Patients who have used anti-CD20 antibody including rituximab (genetical recombination) prior to the informed consent for idiopathic membranous nephropathy
4. Patients who have participated in another clinical study within 12 weeks prior to the informed consent (enrollment is allowed for those participating in a clinical study in the range of 'Indications' or 'Dosage and Administration' in Japan) or patients who are participating in another study
5. Patients with history of renal transplant
6. Patients with poorly controlled diabetes (HbA1c of 8.0% or higher)
7. Patients who have or are suspected to have active infection (infection requiring treatment with systemic antimicrobial, antifungal, or antiviral agents) at the time of informed consent
8. Patients tested positive for HBs antigen, HBs antibody, HBc antibody, and/or HCV antibody (patients with positive HBs antibody and/or HBc antibody can be enrolled only when HBV-DNA test is negative [less than the detection limit]), or patients with positive HIV antibody or HTLV-1 antibody at the time of the screening
9. Patients with leukopenia (less than 2,000 /mm3), neutropenia (less than 1,000 /mm3), or lymphopenia (less than 500 /mm3) at the time of the screening
10. Patients with history of serious hypersensitivity or anaphylactic reaction to one of the ingredients in the investigational drug or murine protein-containing products
11. Patients who are judged to be life-threatening nephrotic syndrome by the investigator or a subinvestigator
12. Patients with serious comorbidity (e.g., hepatic, renal (excluding idiopathic membranous nephropathy with nephrotic syndrome), cardiac, lung, hematologic, or brain disease)
13. Female patients who are pregnant, lactating, or potentially pregnant, patients who are not willing to use contraceptive measures during the study period, or female patients not willing to use contraceptive measures until 12 months after the last dose of study drug (except for female patients who are unale to pregnant)
14. Patients who are judged to be unsuitable by the investigator or a subinvestigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving ICR I | up to 26 weeks
  Achieving ICR I is defined as "Urine protein-creatinine ratio < 1.0 g/gCr".

SECONDARY OUTCOMES:
Percentage of patients who are CR, ICR I, ICR II, NR or PR | up to 26 weeks
  CR, ICR I, ICR II, NR or PR are defied as below; CR (Complete Remission): Urine protein-creatinine ratio < 0.3 g/gCr ICR I (Incomplete Remission Type I): 0.3 g/gCr ≤ Urine protein-creatinine ratio < 1.0 g/gCr ICR II (Incomplete Remission Type II): 1.0 g/gCr ≤ Urine protein-creatinine ratio < 3.5 g/gCr NR (No Response): 3.5 g/gCr ≤ Urine protein-creatinine ratio PR (Partial Remission): Decrease in urine protein-creatinine ratio from base line ≥50%, and urine protein-creatinine ratio 0.3 to 3.5 g/gCr
Duration before achieving CR, ICR I, ICR II or PR | up to 26 weeks
  Duration of achieving CR, ICR I, ICR II or PR is summarized.
Urine protein-creatinine ratio | up to 26 weeks
  The differences of urine protein-creatinine ratio between prior to treatment and at each timepoint are summarized.
eGFR | up to 26 weeks
  The differences of eGFR between prior to treatment and at each timepoint are summarized.
B-cells (CD19-positive and CD20-positive cells) | up to 26 weeks
  B cell counts (CD19 positive and CD20 positive cell counts) at each timepoint are summarized.
Expression of HACA | up to 26 weeks
  The number of patients expressing HACA, and the proportion of these patients at each timepoint are summarized.
Serum rituximab (genetical recombination) concentration | up to 26 weeks
  Serum rituximab (genetical recombination) level at each timepoint are summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Shoichi Shoichi, PhD, MD, Principal Investigator — Nagoya University Hospital
Locations (18):
- Japan (18):
  - Anjo Kosei Hospital, Anjo, Aichi-ken
  - Kasugai Municipal Hospital, Kasugai, Aichi-ken
  - Konan Kosei Hospital, Kōnan, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University hospital, Toyoake, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospial, Kurume, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospial, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Tazuke Kofukai, Medical Research Institute, Kitano Hospital, Osaka, Osaka
  - Osaka University Hospital, Osaka, Osaka
  - Hamamatsu University Hosptial, Hamamatsu, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
If the principal investigator, clinical trial office, main stakeholder conclude that secondary use of individual data obtained in this clinical trial is beneficial for additional analysis, the secondary use of data excluding personal information will be acceptable after publication of results.

REFERENCES:
- [Derived] Shimizu S, Tanaka A, Matsuyama N, Kinoshita F, Furuhashi K, Maruyama S; PRIME Study Group. Randomised, double-blind study to evaluate the efficacy of rituximab in the treatment of idiopathic membranous nephropathy: A clinical trial protocol. PLoS One. 2025 Mar 18;20(3):e0320070. doi: 10.1371/journal.pone.0320070. eCollection 2025. PMID 40100934
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526